CLINICAL TRIAL: NCT03637530
Title: A Prospective Randomized Study of Effect if Lung Protective Ventilation by Reducing Airway Pressure During Laparoscopic Surgery
Brief Title: a Study Conducted About a New Mode of Ventilation in Laparoscopic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences, Rishikesh (Other Government)
Responsible Party: Principal Investigator, ADABALA VIJAY BABU, post graduate,department of Anesthesiology,AIIMS Rishikesh, All India Institute of Medical Sciences, Rishikesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Lung Injury, Acute
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): in this group of patients, inverse ratio ventilation is provided during general anaesthesia
  Interventions: Other: inverse ratio ventilation
- control group (No Intervention): in this group of patients, conventional ventilation is provided during general anaesthesia

INTERVENTIONS:
Other: inverse ratio ventilation — during general anaesthesia in laparoscopic surgeries, this group of patients will receive inverse ratio ventilation with proper observation of hemodynamics
  Arms: intervention group

SUMMARY:
Carbon dioxide insufflations of abdomen are integral part of laparoscopic operations in minimally invasive surgery era. It does cause splinting effect on diaphragm movement and set it high inside thoracic cavity too. In turn it will be associated with increase in peak and plateau airway pressure during positive pressure ventilation. Inverse ratio ventilation has been shown to improve lung compliance and restrict the peak and plateau airway pressure and should be useful as one of the lung protective ventilation method to improve respiratory outcome in laparoscopy surgery.

DETAILED DESCRIPTION:
Anaesthesiologists have been ventilating patients in the perioperative period with relatively large tidal volumes (10-15 ml/kg ideal body weight) to prevent intraoperative atelectasis. Ventilating patient with large tidal volumes may be a risk factor for development of lung injury.During surgical procedures, both general anesthesia and high tidal volumes may strain non injured lungs and trigger inflammation. High tidal volumes that cause alveolar overstretching can contribute to extra pulmonary organ dysfunction through systemic release of inflammatory mediators.

Recently protective lung ventilation strategies has been reported to be useful to reduce the respiratory complications in postoperative period. The use of small tidal volume (Vt), positive end-expiratory pressure (PEEP) and restricting peak airway pressure have shown reduced incidence of ventilation induced lung injury.

It has been shown that a small tidal volume (VT) and PEEP can reduce the incidence of postoperative lung dysfunction and improve intraoperative oxygenation. Restricting peak airway pressure can be achieved by inverse ratio ventilation. Minimizing the risk of ventilator-induced lung injury (VILI), improving oxygenation and alveolar recruitment are all advantages of inverse ratio ventilation. However, the potential utility of pressure controlled inverse ratio ventilation (PCIRV) has not been studied in patients undergoing general anaesthesia.

Investigators hypothesized that in patients with normal lungs scheduled for general anesthesia, PIV might prevent lung function deterioration and lung morphological alterations. Investiagators aim was to compare the intraoperative protective ventilation strategies on oxygenation/ ventilation and postoperative lung dysfunction and lung injury among patients undergoing laparoscopic upper abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* ASA- I and II
* Patients undergoing laparoscopic upper abdominal surgery

Exclusion Criteria:

* Significant pulmonary disease
* Significant cardiac dysfunction
* BMI>30 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
change in partial pressure of oxygen from baseline | upto 1 day postoperatively
  Investigators assume that in laparoscopic surgeries inverse ratio ventilation can be used to decrease the airway pressures

SECONDARY OUTCOMES:
changes in pulmonary function tests from baseline | upto 3 days postoperatively
  Investigators assume that the pulmonary function tests will be improved as we ventilate with inverse ratio ventilation as a protective lung strategy

CONTACTS AND LOCATIONS:
Overall Officials: MUKESH TRIPATHI, MD, Study Director — PROFESSOR AND HOD, ANAESTHESIOLOGY,AIIMS RISHIKESH

IPD SHARING:
Plan to Share IPD: Undecided
I would like to share the results of my trail once it gets completed so that the effectiveness of the intervention will be known to others

REFERENCES:
- [Background] 8. Wang, X.Q., Wang, P.M., Wang, K.G., Jiang, T. and Xu, Z. Pressure-Controlled Inverse Ratio Ventilation during General Anesthesia for Open Abdominal Surgery Improves Postoperative Pulmonary Function. J. Biomedical Science and Engineering, 9, 17-24